CLINICAL TRIAL: NCT04521543
Title: Laparoscopic Sleeve Gastrectomy Under General Anesthesia in Severely Obese Patients: a Single-centered Retrospective Study in China
Brief Title: Laparoscopic Sleeve Gastrectomy Under General Anesthesia in Severely Obese Patients: a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Shengjin Ge,MD, Professor of Anesthesiology, Fudan University
Other Study IDs: B2020-190
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: severely obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the improvement of living standards and changes in living habits in China, obesity has become an important issue. The latest data show that the number of obese people in China has exceeded 100 million. Laparoscopic sleeve gastrectomy (LSG), which reduces the volume of the stomach and maintains the original anatomical structure of the gastrointestinal tract, has been widely used in weight loss surgery for obese patients to improve glucose metabolism and other metabolic disease comorbidities.Anesthesiologists face specific challenges for obese patients: difficult venous and airway access and the risk of obesity-related comorbidity.

Since 2015, the investigator's center has performed LSG and gradually formed a multidisciplinary collaboration procedure for the perioperative management of obese patients. This study aims to summarize the clinical characteristics, anesthesia management and outcomes to optimize the perioperative management and accelerate the recovery of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged>18 years
2. American Society of Anesthesiologists (ASA) status I-III
3. receiving selective laparoscopic sleeve gastrectomy (LSG) under general anesthesia

Exclusion Criteria:

1.BMI<35 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely obese patients underwent laparoscopic sleeve gastrectomy (LSG) under general anesthesia with multidisciplinary collaboration.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The rate of one-time intubation success | during the anesthesia
  the intubation was performed once successfully

SECONDARY OUTCOMES:
number of participants with anesthesia-related complications | Perioperative period
  such as difficult ventilation, difficult intubation, or hoarseness.
the hospital stay (days) | Perioperative period
  total time of hospital stay (days)
the hospitalization cost（Yuan） | Perioperative period
  the total cost of the hospitalization （Yuan）

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China